CLINICAL TRIAL: NCT00022893
Title: Retreatment Study of Patients With Non-Hodgkin's Lymphoma Who Have Previously Responded to Iodine-131 Anti-B1 Antibody.
Brief Title: Safety and Efficacy Study of Iodine-131 Anti-B1 Antibody for the Retreatment of Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Corixa Corporation (Industry)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-98-021
Record Dates: First submitted 2001-08-15; First posted 2001-08-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-08

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Radioimmunotherapy; Monoclonal Antibody; Corixa; Bexxar; Anti-B1 Antibody; Tositumomab; Iodine -131 Anti-B1 Antibody; Iodine I 131 Tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

INTERVENTIONS:
Drug: Iodine-131 Anti-B1 Antibody

SUMMARY:
The purpose of this study is to enable retreatment with Iodine-131 Anti-B1 Antibody therapy for patients with non-Hodgkin's lymphoma (NHL) who previously responded (PR, CCR, or CR) for at least 3 months to Iodine-131 Anti-B1 Antibody therapy.

DETAILED DESCRIPTION:
The endpoints of the study are to determine the response rate, complete response rate, duration of response, time to progression, time-to-treatment failure, safety, and survival following Iodine-131 Anti-B1 Antibody therapy in patients with NHL who previously responded (PR, CCR, or CR) with a duration of response of at least 3 months to Iodine-131 Anti-B1 Antibody therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed initial diagnosis of non-Hodgkin's B-cell lymphoma.
* Patients must have previously responded (PR, CCR, or CR) with a duration of response of at least 3 months to Iodine-131 Anti-B1 Antibody therapy. The patient's disease must have progressed following the response to Iodine-131 Anti-B1 Antibody therapy.
* Patients must have evidence that their tumor tissue expresses the CD20 antigen.
* Patients must have a performance status of at least 60% on the Karnofsky Scale and an anticipated survival of at least 3 months.
* Patients must have an absolute granulocyte count (ANC)>1,500 cells/mm3 (US) or >1,500 x 109/l (UK) and a platelet count >100,000 cells/mm3 (US) or >100,000 x 109/l (UK) within 14 days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine <1.5 x upper limit of normal) and hepatic function (defined as total bilirubin <1.5 x upper limit of normal and hepatic transaminases [AST and ALT] <5 x upper limit of normal) within 14 days of study entry.
* Patients must have bi-dimensionally measurable disease. At least one lesion must be greater than or equal to 2 x 2 cm (by CT scan).

Exclusion Criteria:

* Patients with more than an average of 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 42 days of study entry. Bilateral posterior iliac crest core biopsies are required if the percentage of intratrabecular space involved exceeds 10% on a unilateral biopsy. The mean of bilateral biopsies must be no more than 25%.
* Patients who have received cytotoxic chemotherapy, radiation therapy, immunosuppressants, or cytokine treatment within 4 weeks prior to study entry (6 weeks for nitrosourea compounds) or who exhibit persistent clinical evidence of toxicity. The use of systemic steroids must be discontinued at least 1 week prior to study entry.
* Patients with active obstructive hydronephrosis.
* Patients with evidence of active infection requiring IV antibiotics at the time of study entry.
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years. Patients who have been disease-free of another cancer for greater than 5 years must be carefully assessed at the time of study entry to rule out recurrent disease.
* Patients with known HIV infection.
* Patients with known brain or leptomeningeal metastases.
* Patients who are pregnant or nursing (breastfeeding). Patients of childbearing potential must undergo a serum pregnancy test within 7 days prior to study entry. Males and females must agree to use effective contraception for 6 months following treatment.
* Patients with previous allergic reactions to iodine. This does not include reacting to IV iodine-containing contrast materials.
* Patients with progressive disease within 1 year of irradiation arising in a field that has been previously irradiated with >3500 cGy.
* Patients who became HAMA positive following Iodine-131 Anti-B1 Antibody therapy or patients who are HAMA positive at the time of enrollment.
* Patients who are concurrently receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Stanford University Medical Center, Palo Alto, California
  - Rush Medical Center, Chicago, Illinois
  - University of Michigan Cancer & Geriatric Center, Ann Arbor, Michigan
  - Cornell Medical Center, New York, New York
- Christie Hospital NHS Trust, Manchester, United Kingdom